CLINICAL TRIAL: NCT01988285
Title: Risk Factors and Biomarkers for Diagnosis and Treatment of EoE
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-1122
Record Dates: First submitted 2013-10-25; First posted 2013-11-20 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: Esophagitis; Eosinophilic Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — Specimen Handling; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Esophageal, gastric, and duodenal biopsies, blood samples, saliva, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dysphagia and GERD controls: The cross-sectional arm will consist of patients who are having a clinically indicated endoscopy for reflux and/or dysphagia.
  Cross-sectional participants will have specimens collected and complete a questionnaire.
  Interventions: Other: Specimen Collection; Other: Questionnaires
- Prospective Longitudinal EoE Cases: The prospective longitudinal group will be subjects who have a positive EoE diagnosis during initial endoscopy. This prospective group will be followed up at their clinically indicated endoscopy after their standard of care clinical therapy of swallowed steroids.
  Prospective longitudinal participants will have specimens collected and complete questionnaires s prior to their standard of care clinical therapy of swallowed steroids and at their clinically indicated follow up upper endoscopy.
  Interventions: Other: Specimen Collection; Other: Questionnaires

INTERVENTIONS:
Other: Specimen Collection — Blood collection, possible saliva collection, possible urine collection, and biopsy collection
Other: Questionnaires — Subjects will complete a questionnaire utilizing validated symptom-specific instruments (Mayo Dysphagia Scale; GERD-HRQL Scale). The questionnaire will also record patient demographics, medical history, and current and past medication use

SUMMARY:
Purpose: To validate our previously developed model of risk factors for diagnosis of eosinophilic esophagitis (EoE), and to assess the utility of serum levels of biomarkers in diagnosis and monitoring of treatment of EoE. Participants: Up to a total of 800 participants (approximately 400 with EoE and 400 without EoE) who are referred for upper endoscopy. Procedures: This is a prospective cohort study. Patients will be compared with newly diagnosed EoE to non-EoE controls, obtain baseline measures, reassess EoE patients after treatment, and also reassess untreated controls. Data collection will include questionnaire results, blood collection, and tissue collection (esophageal biopsies performed during upper endoscopy per pre-specified protocol). Blood will be analyzed for the presence of the candidate biomarkers. Patients will be compared with newly diagnosed EoE to non-EoE controls, obtain baseline measures, reassess EoE patients after treatment, and also reassess untreated controls. Data collection will include questionnaire results, blood collection, possible saliva collection, possible urine collection, and tissue collection (esophageal biopsies performed during upper endoscopy per pre-specified protocol). Blood will be analyzed for the presence of the candidate biomarkers, including eotaxin-3 and IL-13.

ELIGIBILITY:
Inclusion Criteria:

1. Referral for upper endoscopy (esophagogastroduodenoscopy; EGD) to evaluate specific symptoms (dysphagia, heartburn, reflux, chest pain, regurgitation, abdominal pain, nausea, or vomiting).
2. Age 18 or older

Exclusion Criteria:

1. Acute GI bleeding.
2. Known cancer of the esophagus, stomach, or small bowel.
3. Prior esophageal resection.
4. Esophageal varices.
5. Active anticoagulation or bleeding diathesis.
6. Medical instability (determined by the performing endoscopist) to precludes performing EGD.
7. Pregnancy
8. Inability to read or understand the consent form and questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of the study population will be patients aged 18 or older presenting at the gastrointestinal (Gl) Endoscopy Clinic at UNC-Chapel Hill for elective upper endoscopy with dysphagia and/or reflux symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Risk factors in EoE diagnosis | Enrollment (day 1)
  To validate our model of clinical, endoscopic, and histopathologic risk factors for diagnosis of EoE by calculating the EoE risk score which includes subject's age, allergic conditions, endoscopic findings, and eosinophil count. Subject's EoE risk scores will be compared between EoE patients and two non-EoE control groups: patients with dysphagia and patients with gastroesophageal reflux disease (GERD) who are not responsive to proton pump inhibitor (PPI) therapy.

SECONDARY OUTCOMES:
Inflammatory serum biomarker measures | Enrollment (day 1)
  To assess operating characteristics of serum biomarkers eotaxin-3 and IL-13 for diagnosis of incident cases of EoE as compared with two non-EoE control groups: patients with dysphagia and patients with GERD who are not responsive to PPI therapy.

OTHER OUTCOMES:
Serum biomarker change following treatment in EoE cases | Enrollment (Day 1) and approximately 8 weeks after initial EGD
  To determine the effect of clinically indicated topical steroid therapy on non-invasive serum biomarkers eotaxin-3 and IL-13 for monitoring treatment response in incident EoE cases.

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No